## CONSENT FORM FOR PARTICIPANTS IN RESEARCH PROJECTS





Title of project: Assessment Of The Volumetric Occlusal Adjustments Required For Michigan Splints Fabricated Using Various Digital Bite Registrations. Version number: 13/07/2024 Ethical review reference number: 43439 Tick or initial 1. I confirm that I have read and understood the information sheet dated (13/07/2024) version 2 for the above project. I have had the opportunity to consider the information and asked questions which have been answered to my satisfaction. 2. I consent voluntarily to be a participant in this project and understand that I can refuse to take part and can withdraw from the project at any time, without having to give a reason. 3. I consent that I have regular dental checks with my dentist and I do not have any current active dental issue. 4. I understand my personal information will be processed for the purposes explained to me in the Information Sheet. I understand that such information will be handled under the terms of UK data protection law, including the UK General Data Protection Regulation (UK GDPR) and the Data Protection Act 2018. 5. I understand that my information may be subject to review by responsible individuals from the College for monitoring and audit purposes. 6. I understand that confidentiality and anonymity will be maintained, and it will not be possible to identify me in any research outputs 7. I agree that the research team can archive my anonymous data for future research projects. 8. I agree that the research team may access my scanned data of the occlusal splints that were fabricated for me records for the purposes of this research project. 9. I understand that I must not take part if I fall under the exclusion criteria as detailed in the information sheet and explained to me by the researcher. 10. I understand that the information I have submitted will be published as a report 11. I consent to my non-identifiable data being stored at a third party data storage provider, [dental lab], as described in the information sheet.

| 12. I consent that I canno the second clinical vis | | the project if the records(scans) were taken at |
|---|---|---|
| Name of Participant | <br>Date | Signature |
| Arwa Alhusban | | Aw |
| Name of Researcher | Date | Signature |